CLINICAL TRIAL: NCT00073294
Title: Phenotypic Assessment of Insulin Resistance and Insulin Secretory Capacity
Brief Title: Insulin Resistance and Insulin Secretion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was not funded
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 9777 (completed)
Record Dates: First submitted 2003-11-18; First posted 2003-11-20 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Diet

INTERVENTIONS:
Behavioral: diet

SUMMARY:
This is a pilot study to examine the prevalence of metabolic risk factors (impaired insulin release and impaired insulin sensitivity) for type 2 diabetes mellitus in children and adults from a population that is at high risk for this disease. We hypothesize that at least one of these pre-diabetic traits will be evident in a large proportion of relatives of known type 2 diabetic children as compared to a control group of subjects without a family history of type 2 diabetes. By isolating these traits, it will be possible to determine the relative contributions of genes and environment to each trait and to identify those at risk for subsequent development of type 2 diabetes by virtue of having one trait. Ultimately, those individuals at risk, especially those with impaired insulin release, would hopefully benefit from intervention to prevent the weight gain that will 'unmask' their underlying pancreatic dysfunction and thus prevent or retard the development of type 2 diabetes.

ELIGIBILITY:
Ascertainment criteria for probands:

* age 10-20 years and
* obesity (BMI >85% for sex and age)
* diabetic criteria as described above or family history (first or second degree relative) with type 2 diabetes

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Columbia Presbyterian Medical Center/ Irving Center, New York, New York
  - Russ Berrie Pavilion, New York, New York